CLINICAL TRIAL: NCT02727972
Title: Examination of Glutamate and mGluR5 in Psychiatric Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1101007933
Record Dates: First submitted 2016-03-17; First posted 2016-04-05 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder; Post-Traumatic Stress Disorder; Bipolar Disorder
Keywords: depression; bipolar; post-traumatic stress disorder; mood disorders; PET; mGluRr; glutamate system; MRI
MeSH Terms: conditions — Depressive Disorder, Major; Stress Disorders, Post-Traumatic; Bipolar Disorder; Depression; Mood Disorders | interventions — Neuropsychological Tests; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Testing (Other): Cognitive assessments
  Interventions: Behavioral: Cognitive Testing
- Magnetic Resonance Imaging (Active Comparator): All subjects will have one MRI with a possibility of one functional MRI (fmri).
  Interventions: Other: MRI
- Positron Emission Tomography (Active Comparator): All subjects will have PET scan using FPEB or ABP688.
  Interventions: Radiation: PET

INTERVENTIONS:
Behavioral: Cognitive Testing — Verbal assessments as well as computer testing.
  Arms: Cognitive Testing
Other: MRI — Anatomical MRIs will be performed on a Siemens 3T Trio at Yale. MR acquisition will be a Sag 3D magnetization-prepared rapid gradient-echo (MPRAGE) sequence with 3.34 ms echo time, 2,500 ms repetition time, 1,000 ms inversion time, 7 degree flip angle, and 180 Hz/pixel bandwidth. The image dimensions will be 256 x 256 x 176 and pixel size 0.98 x 0.98 x 1.0 mm. Resting state MRIs will also be obtained as follows: We will be doing 2 six minute scans with subjects in the scanner, eyes open, fixating a cross. TR = 3 secs 45 slices x 3 mm slice thickness = 13.5 cm. In plane resolution = 3 x 3 mm, slice acquisition order = ascending.
  Other Names: Magnetic Resonance Imaging
  Arms: Magnetic Resonance Imaging
Radiation: PET — High Resolution Research Tomograph (HRRT), the highest resolution human brain scanner available, or HR+ will be used to image subjects. Vital signs (blood pressure, pulse, respiration) will be obtained before and after radiotracer administration. An antecubital venous catheter will be used for IV administration of the radiotracer and for venous blood sampling. A radial artery catheter will be inserted by an experienced physician before the PET scan. At the beginning of each scan, the subject's head will be immobilized and a 6 minute transmission scan using an orbiting 137Cs (HRRT) or 68GE (HR+) point-source is obtained and used for attenuation correction. PET scans will be acquired using bolus or bolus plus constant infusion administration of FPEB or ABP688.
  Other Names: Positron Emission Tomography
  Arms: Positron Emission Tomography

SUMMARY:
This research study is designed to look at the involvement of the glutamate system in depression. Each subject will undergo a screening appointment to determine study eligibility. Thereafter, the study will take 2 or 3 visits depending on schedule availability and will consist of one MRI scan, and PET scan. Subjects will also participate in cognitive testing. Depending on camera time, staff availability and subject schedule, total study participation may last 1-2 months.

DETAILED DESCRIPTION:
With the recent advancements in positron emission tomography (PET) and radioligand development, the investigators are now able to image and quantify the metabotropic glutamatergic system (mGluR5) in vivo in human subjects. The study proposes a novel investigation of mGluR5 in depression to obtain critical data to advance understanding of the etiology of depression and its associated symptoms of cognitive dysfunction.

Aim 1: To determine mGluR5 availability in individuals with mood disorders compared to healthy controls as measured with PET brain imaging.

Hypothesis 1: The study hypothesizes a decrease in mGluR5 availability in individuals with mood disorders in regions responsible for emotional and cognitive processes, including the amygdala, hippocampus, thalamus, anterior cingulate, and frontal cortices.

Aim 2: To determine if glutamate cycling in individuals with mood disorders is altered as compared to healthy controls as measured with [1H]MRS and [13C]MRS.

Hypothesis 2: The study hypothesizes an increase in glutamate number in individuals with mood disorders as compared to controls.

Aim 3: To determine if the PET alterations in the glutamatergic system of depressed individuals are associated with cognitive deficits observed in depression, including concentration, attention, memory, distractibility, and startle.

Hypothesis 3: The study hypothesizes a positive relationship between mGluR5 availability and cognitive functioning, such that individuals with higher receptor availability will perform better on tests of concentration, attention, memory, distractibility, and startle than individuals with lower receptor availability.

Aim 4: To determine mGluR5 availability in individuals with anxiety and schizophrenia compared to healthy controls as measured with PET brain imaging.

Hypothesis 4: Anxiety disorders such as obsessive compulsive disorder, and delusional disorders such as schizophrenia are frequently comorbid with mood disorders, and the glutamatergic system has been observed to be compromised in these individuals as well. This study will examine if there are regional differences in mGluR5 availability between individuals with depression, bipolar disorder, obsessive compulsive disorder, and schizophrenia.

Aim 5: To examine whether changes in mGluR5 availability are dependent on state, or whether the lower availability is due to trait.

Hypothesis 5: Due to changes in endogenous GLU shown with MRS studies, this study hypothesizes normalization (or increase) in mGluR5 availability in euthymia as compared to depressed state.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* Subjects will be between the ages of 18-70 years old
* English speaking
* No other DSM-5 diagnosis present, besides required as below

Inclusion criteria for acute depressed subjects:

* Clinical diagnosis of a current depressive episode
* Medication-free for at least 2 weeks or medicated with a permissible medication

Inclusion criteria for PTSD subjects:

* Clinical diagnosis of current PTSD as per DSM-5
* Medication free for at least 2 weeks or medicated with a permissible medication

Inclusion criteria for healthy controls:

* No current, or history of, any DSM-5 diagnosis

Exclusion Criteria:

* Have a current or past significant medical, neurological or metabolic disorder or head injury that lead to significant long term decline in cognitive abilities as seen by decline in grades or work performance
* Have significant medical illness such that would contraindicate study participation based on above criteria and PI/MD history review
* Have active, significant suicidal ideation
* Have implanted metallic devices or any MR contraindications
* Are women who are pregnant or breastfeeding
* Met DSM-5 criteria for mild substance use disorder (except nicotine and marijuana) within the past 6 months or met DSM-5 criteria for moderate to severe substance use disorder (except nicotine and marijuana) within the past year
* Have history of prior radiation exposure for research purposes within the past year such that participation in this study would place them over FDA limits for annual radiation exposure. This guideline is an effective dose of 5 rem received per year
* Have given a blood donation within eight weeks of the start of the study
* Have history of a bleeding disorder or are currently taking anticoagulants (such as Coumadin, Heparin, Pradaxa, Xarelto)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-02-21 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Evidence of glutamate availability (mGluR5) in psychiatric disorders confirmed by MRI and PET data. | Through study completion date, an average of 4 years.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Esterlis, PhD, Principal Investigator — Yale University
Locations (1):
- PET Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No